CLINICAL TRIAL: NCT07030894
Title: A Prospective, Single-Arm Clinical Study of Budesonide in Combination With Ambrisentan for the Treatment of Patients With IgA Nephropathy
Brief Title: Nefecon and Ambrisentan in IgA Nephropathy
Acronym: BAIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25K183-001
Record Dates: First submitted 2025-06-08; First posted 2025-06-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: IgA Nephropathy; Chronic Kidney Disease; Proteinuria
Keywords: Proteinuria; IgA Nephropathy; Budesonide; Ambrisentan; Single-arm trial
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy (Experimental): Subjects who meet the screening criteria will be treated with Budesonide in combination with Ambrisentan. Budesonide , 16mg/d for 36 weeks, taken orally. Ambrisentan , 5mg/d for 36 weeks, taken orally.
  Interventions: Drug: "Nefecon®","Ambrisentan"

INTERVENTIONS:
Drug: "Nefecon®","Ambrisentan" — Subjects who meet the screening criteria will be treated with Budesonide in combination with Ambrisentan.
  Budesonide (Nefecon®), 16mg/d for 36 weeks, taken orally. Ambrisentan , 5mg/d for 36 weeks, taken orally.

SUMMARY:
Application of Budesonide in Combination with Ambrisentan in the treatment of IgA nephropathy with progression ESKD risk (24-hour urinary protein ≥ 0.5g/24h), observing the degree and safety of reducing urinary protein and delaying eGFR progression, and observing changes in serum Gd-IgA1 levels

DETAILED DESCRIPTION:
This study is a prospective, single arm clinical trial planned to recruit 129 patients with primary IgA nephropathy. Including a screening period and a treatment period, a total of 6 visits were conducted. The screening period was completed within 30 days before the treatment period, and the medical history, medication, and examination results collected during the visits were used as the basis for screening subjects in this study. Subjects who met the inclusion criteria but did not meet any exclusion criteria were enrolled in the study and treated with Budesonide in combination with Ambrisentan for a total of 36 weeks. After the end of the trial, data from 129 enrolled patients were analyzed for statistical analysis. If the treatment is effective, randomized controlled trials will be added to validate it when conditions permit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IgA nephropathy by pathological biopsy within 4 years;
* Age between 18 and 70 years old;
* 0.5g/24h ≤ 24-hour urinary protein;
* The estimated glomerular filtration rate (eGFR) calculated using the CKD-EPI formula satisfies: eGFR ≥ 30 mL/min/1.73 ㎡

Exclusion Criteria:

* Exclude special pathological or clinical kidney disease types such as crescentic glomerulonephritis (pathological diagnosis>50%), minimal change nephropathy with IgA deposition, etc;
* Exclude secondary IgA nephropathy, including allergic purpura, ankylosing spondylitis, systemic lupus erythematosus, Sjogren's syndrome, viral hepatitis, cirrhosis, rheumatoid arthritis, and mixed connective tissue disease;
* Select patients who have experienced any of the following cardiovascular events within the previous 12 weeks: myocardial infarction, unstable angina, ventricular arrhythmia, New York Heart Association class II or above heart failure, stroke, etc;
* Within 12 weeks prior to the first medication, systemic use (excluding local and nasal inhalation use) of immunosuppressants, including but not limited to glucocorticoids, cyclophosphamide, azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, rituximab, Tripterygium wilfordii, etc; Have used an endothelin receptor antagonist within 12 weeks prior to the first medication;
* Active tuberculosis patients and untreated latent tuberculosis patients;
* Patients with active hepatitis or latent hepatitis B (patients with HBcAb positive and HBV DNA positive); According to the results of the five hepatitis B tests, patients with HBsAg positivity should be excluded; Patients who are HBsAg negative but HBcAb positive, regardless of whether HBsAb is positive or negative, need to be tested for HBV-DNA to determine their condition: if HBV-DNA is positive, the patient needs to be excluded; If HBV-DNA is negative, patients can participate in the trial;
* History of immunodeficiency diseases or positive HIV test results (enzyme-linked immunosorbent assay and protein immunoblotting);
* Patients diagnosed with malignant tumors within the past 5 years, except for treated basal cell carcinoma of the skin, effectively resected squamous cell carcinoma of the skin, colon polyps, or cervical cancer in situ;
* Patients undergoing kidney transplantation;
* Pregnant women, lactating women, and men or women with fertility plans during the trial period;
* For individuals allergic to human derived biological products;
* Patients who have received any clinical trial medication within 4 weeks prior to their first use;
* Participants deemed unsuitable by researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in UPCR (24h urine) | From enrollment to the end of treatment at 36 weeks

SECONDARY OUTCOMES:
Change in eGFR | From enrollment to the end of treatment at 36 weeks
Changes in IgA/IgG/IgM and Gd-IgA1 levels at all visits | From enrollment to the end of treatment at 36 weeks
Annualized eGFR slope at Week 36 | From enrollment to the end of treatment at 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China